CLINICAL TRIAL: NCT06258733
Title: Food Literacy Intervention for Arab and Jewish Women in the Jerusalem Region - is a "Train the Trainer" Approach Feasible and Effective?
Brief Title: Food Literacy Intervention - is a "Train the Trainer" Approach Feasible and Effective?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FL-COST-HMO-CTIL
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lifestyle Risk Reduction; Health Behavior; Food Habits
MeSH Terms: conditions — Risk Reduction Behavior; Health Behavior; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study with two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lay-led FL workshops (Experimental): Community lay leaders who underwent training in a manualized program will disseminate the workshop to women in their communities through engaging visual and game-based tools.
  Interventions: Behavioral: Lay-led FL workshops
- Expert-led FL workshops (Experimental): Trained health experts will disseminate the same manualized program in community groups recruited by research staff to match lay-led groups.
  Interventions: Behavioral: Expert-led workshops

INTERVENTIONS:
Behavioral: Lay-led FL workshops — Groups of women recruited by trained lay-leaders will receive an 8-session lay-led FL workshop. Workshop participants will receive a self-report baseline survey at the first session, and post surveys at the last session and 3 months after the last session. The surveys will be anonymous and will be conducted and collected by the lay workshop facilitator. Lay-leaders will receive an incentive to collect surveys from workshop participants. A member of the research staff will be present at the time of the survey collection to ensure data are collected according to protocol. Monthly phone calls with lay-leaders will take place to ensure implementation in the community, including problem solving and help maintaining motivation. To help ensure implementation in the lay-led arm, lay leaders will be required to complete one workshop in the community before receiving a graduation certificate.
  Arms: Lay-led FL workshops
Behavioral: Expert-led workshops — Matching groups of women recruited by research staff will receive the same 8-session expert-led FL workshop. Workshop participants will receive a self-report baseline survey at the first session, and post surveys at the last session and 3 months after the last session. The surveys will be anonymous and will be conducted and collected by the expert workshop facilitator.
  Arms: Expert-led FL workshops

SUMMARY:
Food literacy (FL) is the capability to make healthy food choices in different contexts, settings and situations. Although eating habits are shaped by different circumstances and skills, most nutrition programs focus on nutrition knowledge alone. Addressing factors such as competencies, self-efficacy and social norms enables sustainable positive change in nutrition behaviour. This study will assess a lay leader-led FL workshop to Arab and Jewish women from disadvantaged communities in the Jerusalem region, utilizing a train-the-trainer approach, and will compare the effectiveness and cost-effectiveness of a lay-led FL intervention to an expert-led intervention.

DETAILED DESCRIPTION:
Food literacy (FL) is the capability to make healthy food choices in different contexts, settings and situations. Although eating habits are shaped by different circumstances and skills, most nutrition programs focus on nutrition knowledge alone. Addressing factors such as competencies, self-efficacy and social norms enables sustainable positive change in nutrition behaviour. This study will assess a lay leader-led FL workshop to Arab and Jewish women from disadvantaged communities in the Jerusalem region, utilizing a train-the-trainer approach, and will compare the effectiveness and cost-effectiveness of a manualized FL intervention given by trained lay-leaders vs. the same workshop given by experts.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew or Arabic literate women who are over 25 years old

Exclusion Criteria:

* Women who do not meet inclusion criteria.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in the effectiveness in raising FL level of a FL workshop given by trained lay leaders vs. experts | At baseline, last workshop session- up to five weeks since baseline, and three months after intervention
  Level of food literacy will be assessed by using a the validated Modified Self-Perceived Food Literacy Scale (M-SPFL) , including 23 questions, mean score ranging between 1-5, the higher the score the higher the food literacy level.
Cost-effectiveness ratio of a FL workshop led by trained lay leaders vs. experts | After 16 workshops in each arm are implemented. Approximately one year after the beginning of the study.
  Cost-effectiveness analysis will compare the two alternatives by calculating the incremental Cost-Effectiveness Ratio (ICER). The Markov chain model will be used to predict short and long-term costs and effectiveness in both arms.

SECONDARY OUTCOMES:
Change in Mediterranean Diet adherence | At baseline, last workshop session- up to five weeks since baseline, and three months after intervention
  Level of adherence to the Mediterranean Diet will be assessed by the Israeli Mediterranean Diet Adherence Screener (I-MEDAS) self-report validated scale. The scale includes 17 items, score ranging between 1-17, the higher the score the higher the food literacy level.

CONTACTS AND LOCATIONS:
Overall Officials: Donna R Zwas, MD, MPH, Principal Investigator — Hadassah Medical Organization; Yael Bar-Zeev, MD, MPH, PhD, Principal Investigator — Hebrew University of Jerusalem

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greenberg KL, Zwas DR, Donchin M, Bar-Zeev Y. Validation and adaptation of the self-perceived food literacy scale (SPFL) among Hebrew and Arabic speaking women in Israel. BMC Public Health. 2025 Dec 4;26(1):124. doi: 10.1186/s12889-025-25597-6. PMID 41339836
- [Background] Artinian NT, Fletcher GF, Mozaffarian D, Kris-Etherton P, Van Horn L, Lichtenstein AH, Kumanyika S, Kraus WE, Fleg JL, Redeker NS, Meininger JC, Banks J, Stuart-Shor EM, Fletcher BJ, Miller TD, Hughes S, Braun LT, Kopin LA, Berra K, Hayman LL, Ewing LJ, Ades PA, Durstine JL, Houston-Miller N, Burke LE; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing. Interventions to promote physical activity and dietary lifestyle changes for cardiovascular risk factor reduction in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 27;122(4):406-41. doi: 10.1161/CIR.0b013e3181e8edf1. Epub 2010 Jul 12. No abstract available. PMID 20625115
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Kalter-Leibovici O, Chetrit A, Lubin F, Atamna A, Alpert G, Ziv A, Abu-Saad K, Murad H, Eilat-Adar S, Goldbourt U. Adult-onset diabetes among Arabs and Jews in Israel: a population-based study. Diabet Med. 2012 Jun;29(6):748-54. doi: 10.1111/j.1464-5491.2011.03516.x. PMID 22050554
- [Background] Vidgen HA, Gallegos D. Defining food literacy and its components. Appetite. 2014 May;76:50-9. doi: 10.1016/j.appet.2014.01.010. Epub 2014 Jan 22. PMID 24462490
- [Background] Wang H, Dwyer-Lindgren L, Lofgren KT, Rajaratnam JK, Marcus JR, Levin-Rector A, Levitz CE, Lopez AD, Murray CJ. Age-specific and sex-specific mortality in 187 countries, 1970-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2071-94. doi: 10.1016/S0140-6736(12)61719-X. PMID 23245603
- [Background] Abu-Saad K, Endevelt R, Goldsmith R, Shimony T, Nitsan L, Shahar DR, Keinan-Boker L, Ziv A, Kalter-Leibovici O. Adaptation and predictive utility of a Mediterranean diet screener score. Clin Nutr. 2019 Dec;38(6):2928-2935. doi: 10.1016/j.clnu.2018.12.034. Epub 2019 Jan 5. PMID 30642736
- [Background] Poelman MP, Dijkstra SC, Sponselee H, Kamphuis CBM, Battjes-Fries MCE, Gillebaart M, Seidell JC. Towards the measurement of food literacy with respect to healthy eating: the development and validation of the self perceived food literacy scale among an adult sample in the Netherlands. Int J Behav Nutr Phys Act. 2018 Jun 18;15(1):54. doi: 10.1186/s12966-018-0687-z. PMID 29914503